CLINICAL TRIAL: NCT06811272
Title: A Phase 2 Study of Outpatient Epcoritamab as Second Line Therapy in Non-Transplant Eligible Relapsed/Refractory Large B-cell Lymphoma
Brief Title: Outpatient Epcoritamab as 2L in NTE R/R DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genmab (Industry)
Responsible Party: Principal Investigator, Julie E. Haydu, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-006
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Large B-cell Lymphoma; Refractory Large B-cell Lymphoma
Keywords: Non-Transplant Eligible; Second Line Therapy; DLBCL; HGBCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epcoritamab (Experimental): Epcoritamab will be a subcutaneous injection on cycle 1-3 days 1, 8, 15, and 22, cycle 4-9 days 1 and 15, and cycle 10 and onwards day 1. Participants in a complete response will discontinue epcoritamab therapy after 12 cycles. Participants in a partial response or with stable disease at 1 year will continue epcoritamab and will discontinue at 18 or 24 months if in a complete response by those timepoints, otherwise they will continue until progression or intolerance.
  Dexamethasone (prophylactic corticosteroid) will be given during initial doses of study treatment. Dexamethasone will be taken either once daily or twice daily while receiving epcoritamab. A drug diary will be provided to participants to document information about dexamethasone being taken.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Bispecific IgG1 antibody

SUMMARY:
The purpose of this study is to measure the efficacy of the study drug, epcoritamab, in participants with relapsed/refractory large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a phase 2 study of outpatient administration of epcoritamab in non-transplant eligible large B-cell lymphoma that has relapsed after, or is refractory to, 1 prior line of therapy.

Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has approved epcoritamab as a treatment option for your disease after at least two prior treatments.

The study treatment may continue for up to 24 cycles or until disease progression, unacceptable toxicity, or withdrawal. Participants will be followed for up to 24 months after last dosage of epcoritamab, or until disease progression or withdrawal, whichever occurs first. After 24 months or at time of progression, participants may be followed annually for survival status.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have large B-cell lymphoma of one of the following histologic subtypes by WHO criteria:

  * Diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS)
  * High grade B-cell lymphoma (HGBCL) with rearrangements of MYC and BCL2 and/or BCL6
  * HGBCL NOS
  * EBV+ DLBCL
  * Primary mediastinal B-cell lymphoma
  * T-cell/histiocyte rich LBCL
  * Grade 3B follicular lymphoma
  * Large B-cell lymphoma transformed from underlying indolent NHL
* PET measurable disease per Lugano criteria.
* Relapsed or refractory disease treated with 1 prior systemic antineoplastic line of therapy that includes an anti-CD20 monoclonal antibody and an anthracycline or an alkylating agent. Patients who have received more than 1 prior systemic antineoplastic line of therapy are not eligible.
* Age ≥18 years.
* ECOG performance status 0-2.
* Not a candidate for high dose chemotherapy and autologous stem cell transplant per the treating investigator, or patient refusal of high dose chemotherapy and autologous transplant.
* Participants must meet the following organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL (Growth factor support is permitted)
  * platelets ≥75,000/mcL (>50,000 in the presence of bone marrow involvement or splenomegaly; platelet transfusions are permitted)
  * Hemoglobin ≥8 g/dL (>7 g/dL in the presence of bone marrow involvement; blood transfusions are permitted)
* Participants must have adequate organ function as defined below (unless abnormalities are considered related to target organ involvement or compression by lymphoma):

  * total bilirubin ≤ 1.5x institutional upper limit of normal (ULN) (Isolated bilirubin ≤3.0x ULN is acceptable if considered secondary to Gilbert's syndrome)
  * AST(SGOT) and ALT(SGPT) ≤3.0x institutional ULN
  * Creatinine clearance ≥45 mL/min eGFR (Cockcroft-Gault or MDRD equation)
  * PT within institutional normal range (unless on anticoagulation expected to affect PT, in which case PT cut off does not apply)
  * PTT within institutional normal range (unless on anticoagulation expected to affect PTT, in which case PTT cut off does not apply)
* Ability to remain within 60 minutes of the administration site for 24 hours following cycle 1 day 15 dose of study drug.
* The effects of epcoritamab on the developing human fetus are unknown. Women of child-bearing potential must agree to use adequate contraception starting with the first dose of study drug, for the duration of study participation, and for at least 6 months after the last dose of study intervention. Women must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Adequate contraception methods:

  * Male Partner Sterilization: When the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate.
  * Use of a combination of any two of the following (one from "a" and one from "b"):

    1. Placement of an intrauterine device (IUD) or intrauterine system or established use of oral, injected, or implanted hormonal methods of contraception
    2. Barrier methods of contraception: Male Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
* True abstinence, defined as refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject.
* Nonchildbearing potential is defined as follows:

  * ≥45 years of age and has not had menses for at least 12 consecutive months.
  * Subjects who have been amenorrhoeic for <1 year must have, on at least two occasions prior to first dose of study drug, a follicle stimulating hormone value greater than 40 IU/L; historical follicle stimulating hormone values are eligible
  * Post-bilateral oophorectomy (with or without hysterectomy) or post-tubal ligation at least six weeks prior to first dose of study drug. Documented oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure. In the case of oophorectomy alone, reproductive status must be confirmed by follicle stimulating hormone level assessment as above.
* Women of childbearing potential (WOCBP) must have a negative highly sensitive serum pregnancy test at screening.
* Fertile men, defined as all males physiologically capable of conceiving offspring who are sexually active with a female partner of childbearing potential, must agree to use adequate contraception starting with the first dose of study drug, for the duration of study participation, and 3 months after completion of administration. Men must also agree not to donate sperm during this period. Men may agree to remain abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term or persistent basis) OR agree to use a male condom, and their female partner must use an additional highly effective contraceptive method with a failure rate of <1% per year when having sexual intercourse if they are a WOCBP (including pregnant females).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participant must not have used an investigational drug or approved systemic lymphoma therapy within 28 days preceding the first dose of study drug. Steroids for lymphoma disease control are permitted but must be stopped at least 7 days prior to the first dose of study drug.
* Participants must not have received prior CD20/CD3 bispecific antibody.
* Participants must not have received prior autologous or allogeneic stem cell transplant.
* Participants must not have received prior anti-CD19 CAR T-cell therapy.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia. At the discretion of the overall PI, participants with residual toxicities > Grade 1 may be considered eligible if in the opinion of the overall PI the residual toxicity is not likely to interfere with the safety or efficacy assessment of the investigational regimen. For residual hematologic toxicities greater than Grade 1.
* Participants must not have known central nervous system involvement by lymphoma.
* Participants must not have a current life-threatening illness, medical condition, or organ system dysfunction (other than the disease under study) which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.
* Participants must not have an uncontrolled active infection. Localized fungal infection of skin or nails are permitted.
* Participants must not have active uncontrolled autoimmune disease. Autoimmune disease under control with chronic systemic corticosteroids at a dose of 10 mg/day of prednisone or less, or equivalent corticosteroid, are eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to epcoritamab. A history of an infusion reaction to CD20-directed therapy is not considered an allergic reaction.
* Women who are pregnant are excluded from this study because it is unknown if epcoritamab can cause embryo-fetal harm when administered to a pregnant woman. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with epcoritamab, breastfeeding should be discontinued if the mother is treated with epcoritamab on study.
* Participant must not have active uncontrolled HIV infection. Participants with HIV are eligible if disease is adequately controlled on an antiretroviral regimen that is in accordance with the current international AIDS Society guidelines, with adequate control defined by presence of both an undetectable viral load, a CD4 count >350, no evidence of AIDS-defining illness (with the exception of a lymphoma diagnosis), and no active opportunistic infections (infections controlled on appropriate anti-infective therapy are permitted).
* Participant must not have active hepatitis B infection. Participants with positive HBV core antibody or HBV surface antigen at screening are eligible if HBV viral load is negative by PCR and they are on appropriate antiviral therapy.
* Participant must not have active hepatitis C infection. Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained. Note: Participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* Subject has no known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. If a subject has signs/symptoms suggestive of SARS-CoV-2 infection or has had recent known exposure to someone with SARS-CoV-2 infection, the subject must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection. Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations. Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen after they meet the following SARS-CoV-2 infection viral clearance criteria: No signs/symptoms suggestive of active SARS-CoV-2 infection AND negative testing (molecular (e.g., PCR) result or 2 negative antigen test results at least 24 hours).
* Participants must not have received a live virus vaccine within 28 days of first dose of study drug.
* Participants must not have any known past or current malignancy other than inclusion diagnosis, except for:

  1. Cervical carcinoma of Stage 1B or less.
  2. Non-invasive basal cell or squamous cell skin carcinoma.
  3. Non-invasive, superficial bladder cancer.
  4. Prostate cancer with a current PSA level <0.1 ng/mL.
  5. Any curable cancer with a complete response (CR) of >2 years duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
12-month progression free survival (PFS) | Day 1 until date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 12 months after initial dose of study treatment.
  The time from registration to the earlier of progression or death due to any cause and will be defined as the percent of patients alive and progression-free at 12 months. Participants alive without disease progression are censored at date of last disease evaluation.

SECONDARY OUTCOMES:
Complete Response Rate | Day 1 to 24 months post treatment
  The proportion of subjects achieving an objective response of complete response (CR) according to the Lugano Classification, prior to start of another non-study anticancer therapy.
Overall Response Rate | Day 1 to 24 months post treatment
  The proportion of subjects achieving an objective response of complete response (CR) or partial response (PR) according to the Lugano Classification, prior to start of another non-study anticancer therapy.
Median Duration of Response | Date of first response to first documented disease progression or date of death from any cause, whichever came first, assessed up to 24 months post treatment
  The time from first response to disease progression or death, and will be summarized using Kaplan-Meier estimates.
Median Duration of Complete Response | Date of complete response to first documented disease progression or date of death from any cause, whichever came first, assessed up to 24 months post treatment
  The time subjects achieve complete response to disease progression or death and will be estimated using Kaplan Meier method or cumulative incidence curves.
Overall Survival | Registration date to date of death from any cause or last known alive date, assessed up to 24 months post treatment
  The time from registration to death due to any cause or censored at date last known alive and will be summarized using Kaplan-Meier estimates.
Incidence and Severity of Treatment-Emergent Adverse Events | Day 1 to 24 months post treatment
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All participants will be followed and assessed for safety and tolerability of the protocol therapy.
Median Time to Resolution of Cytokine Release Syndrome | Date of cytokine release syndrome to resolution date of cytokine release syndrome
  The duration of time for subjects to resolve cytokine release syndrome (CRS) and will be estimated using Kaplan Meier method or cumulative incidence curves.
Median Time to Resolution of Immune Effector Cell-Associated Neurotoxicity Syndrome | Date of immune effector cell-associated neurotoxicity syndrome to resolution date of immune effector cell-associated neurotoxicity syndrome
  The duration of time for subjects to resolve immune effector cell-associated neurotoxicity syndrome (ICANS) and will be estimated using Kaplan Meier method or cumulative incidence curves.
Proportion of Subjects Receiving Interventions for CRS and/or ICANS | Date of intervention for CRS and/or ICANs to resolution of CRS and/or ICANS
  The number of subjects receiving interventions for CRS and ICANS, CRS, or ICANS and will be estimated using Kaplan Meier method or cumulative incidence curves.
Rate of Hospitalization | Day 1 to 24 months post treatment
  The frequency of subjects that are hospitalized and will be estimated using Kaplan Meier method or cumulative incidence curves.
Rate of Emergency Room Visits | Day 1 to 24 months post treatment
  The frequency of subjects that go to the emergency room and will be estimated using Kaplan Meier method or cumulative incidence curves.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E. Haydu, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Julie E. Haydu, MD, PhD (julie_haydu@mgh.harvard.edu) at 617-724-4000. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation